CLINICAL TRIAL: NCT05236426
Title: Comparison of Cardiac Index (CI) Measurements Performed With Use of the Bioreactance Technology and Transpulmonary Thermodilution in Reference to Measurements Based on Echocardiography.
Brief Title: Comparison of Cardiac Index (CI) Measurements Performed With Different Methods
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Jan Adamski, Principal Investigator, University of Warmia and Mazury in Olsztyn
Other Study IDs: UWMOlsztyn
Record Dates: First submitted 2022-01-31; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Hemodynamic Instability
Keywords: hemodynamic monitoring; cardiovascular monitoring; bioreactance; echocardiography; pulmonary thermodilution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The aim of the study is to determine the correlation of the results of cardiac index (CI) measurements performed with use of bioreactance technology with the results of measurements made with the use of transpulmonary thermodilution. Both methods will be evaluated in reference to measurements based on echocardiography.

DETAILED DESCRIPTION:
After approval of the study design by the institutional ethics committee, 50 critically ill adult patients (requiring haemodynamic monitoring and mechanical ventilation) treated in the ICU for a intracranial pathology will be enrolled in the study.

Exclusions: Age under 18, presence of pleural effusion or pericardium (confirmed by chest X-ray and / or ultrasound / echocardiography), presence of aortic / mitral valve disease, presence of an implanted pacemaker CI measurements will be performed simultaneously for 5 minutes. The CI value measured by the transpulmonary thermodilution technique will be obtained with the PiCCO system (Pulsiocat PV8115; Pulsion Medical Systems, Feldkirchen, Germany). Measurements will be made three times within 5 minutes. For statistical purposes, the value of the arithmetic mean of the obtained results will be used.

The CI value as measured by the bioreactance method will be determined using the monitor: Starling Fluid Management System (Baxter International Inc, USA). This monitor uses bioreactance technology to determine hemodynamic parameters and bioimpedance technology to measure thoracic fluid content (TFC). The test data will be recorded with two pairs of electrodes placed on the chest according to the manufacturer's instructions. Measurements documented at 30-second intervals will concern 10 measurement cycles. The average of the obtained results will be subjected to statistical analysis.

Echocardiographic examination of the heart to determine the value of CI will be performed by one (always the same) qualified (certified in echocardiographic examinations) clinician.

Echocardiographic measurements will begin with determining the diameter of the left ventricular outflow tract (left ventricular outflow tract cross-sectional area, LVOT-CSA). Then, three subvalvular velocity time integral (LVOT-VTI) measurements will be made over the course of 5 minutes. This measurement will be performed in the apical five-chamber projection.

The stroke volume (SV) value will be calculated as: SV = LVOT-CSA x LVOT-VTI. The CI value will be calculated using the formula: CI = SV x heart rate (HR) / body surface area (BSA). The CI value archived for further statistical analysis will be the average of three measurements performed within 5 minutes.

Other variables that will be documented simultaneously with CI measurements: patient gender and weight, use of vasospastic / inotropic drugs (dose mcg / kg / min), positive end expiratory pressure (PEEP), presence of pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 50 critically ill adult patients (requiring haemodynamic monitoring and mechanical ventilation) treated in the ICU for a intracranial pathology

Exclusion Criteria:

* Age under 18
* Presence of pleural effusion or pericardium (confirmed by chest X-ray and / or ultrasound / echocardiography)
* Presence of aortic / mitral valve pathology
* Presence of an implanted pacemaker

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 critically ill adult patients (requiring haemodynamic monitoring and mechanical ventilation) treated in the ICU for intracranial pathology
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac Index value measured by the transpulmonary thermodilution technique | The results of three measurements will be documented within five minutes
  The cardiac index is expressed with units : Liters/minute/meter2
Cardiac Index value measured with use of bioreactance technology | The results of ten measurements at intervals of 30 seconds will be documented within five minutes
  The cardiac index is expressed with units : Liters/minute/meter2
Cardiac index value determined with use an ultrasound technique (echocardiography) | The results of three measurements will be documented within five minutes
  The cardiac index is expressed with units : Liters/minute/meter2

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Geerts BF, Aarts LP, Jansen JR. Methods in pharmacology: measurement of cardiac output. Br J Clin Pharmacol. 2011 Mar;71(3):316-30. doi: 10.1111/j.1365-2125.2010.03798.x. PMID 21284692
- [Background] Demiselle J, Mercat A, Asfar P. Is there still a place for the Swan-Ganz catheter? Yes. Intensive Care Med. 2018 Jun;44(6):954-956. doi: 10.1007/s00134-018-5158-0. Epub 2018 May 23. No abstract available. PMID 29796915
- [Background] Kobe J, Mishra N, Arya VK, Al-Moustadi W, Nates W, Kumar B. Cardiac output monitoring: Technology and choice. Ann Card Anaesth. 2019 Jan-Mar;22(1):6-17. doi: 10.4103/aca.ACA_41_18. PMID 30648673
- [Background] Keren H, Burkhoff D, Squara P. Evaluation of a noninvasive continuous cardiac output monitoring system based on thoracic bioreactance. Am J Physiol Heart Circ Physiol. 2007 Jul;293(1):H583-9. doi: 10.1152/ajpheart.00195.2007. Epub 2007 Mar 23. PMID 17384132
- [Background] Squara P, Denjean D, Estagnasie P, Brusset A, Dib JC, Dubois C. Noninvasive cardiac output monitoring (NICOM): a clinical validation. Intensive Care Med. 2007 Jul;33(7):1191-1194. doi: 10.1007/s00134-007-0640-0. Epub 2007 Apr 26. PMID 17458538
- [Background] Raval NY, Squara P, Cleman M, Yalamanchili K, Winklmaier M, Burkhoff D. Multicenter evaluation of noninvasive cardiac output measurement by bioreactance technique. J Clin Monit Comput. 2008 Apr;22(2):113-9. doi: 10.1007/s10877-008-9112-5. Epub 2008 Mar 14. PMID 18340540
- [Background] Porter TR, Shillcutt SK, Adams MS, Desjardins G, Glas KE, Olson JJ, Troughton RW. Guidelines for the use of echocardiography as a monitor for therapeutic intervention in adults: a report from the American Society of Echocardiography. J Am Soc Echocardiogr. 2015 Jan;28(1):40-56. doi: 10.1016/j.echo.2014.09.009. No abstract available. PMID 25559474
- [Background] Malik SB, Chen N, Parker RA 3rd, Hsu JY. Transthoracic Echocardiography: Pitfalls and Limitations as Delineated at Cardiac CT and MR Imaging. Radiographics. 2017 Mar-Apr;37(2):383-406. doi: 10.1148/rg.2017160105. Epub 2017 Feb 17. PMID 28212053
- [Background] Ling HZ, Gallardo-Arozena M, Company-Calabuig AM, Nicolaides KH, Kametas NA. Clinical validation of bioreactance for the measurement of cardiac output in pregnancy. Anaesthesia. 2020 Oct;75(10):1307-1313. doi: 10.1111/anae.15110. Epub 2020 May 29. PMID 32469423
- [Background] Lamia B, Kim HK, Severyn DA, Pinsky MR. Cross-comparisons of trending accuracies of continuous cardiac-output measurements: pulse contour analysis, bioreactance, and pulmonary-artery catheter. J Clin Monit Comput. 2018 Feb;32(1):33-43. doi: 10.1007/s10877-017-9983-4. Epub 2017 Feb 10. PMID 28188408